CLINICAL TRIAL: NCT03907254
Title: Biopsychosocial Effect of Service Dog Training on Post-traumatic Stress (PTS) and Post Concussive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-2018-0159
Record Dates: First submitted 2019-03-12; First posted 2019-04-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Post-traumatic Stress Disorder; Posttraumatic Stress Disorder; Traumatic Brain Injury
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Up to 156 participants will be recruited in the National Capital Region (NCR) for a ten-week longitudinal pre-post study, in which each participant will serve as their own control. Additionally, up to 104 participants will be recruited for a three-week longitudinal parallel-randomized study through the National Intrepid Center of Excellence (NICoE) four-week Intensive Outpatient Program (IOP). A three-month post-intervention follow-up will be conducted for both designs (optional for IOP participants).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- National Capital Region (NCR) (Experimental): 10-week longitudinal pre-post study, in which each participant will serve as their own control. Each participant will train a service dog using methods that facilitate a relationship between the trainer and dog for the gradual shaping of desired behavior. Self-report measures of behavioral symptoms will be given weekly throughout participation in this study. Biological measures, including blood collection, HR, BP, etc. will be collected at baseline, during the three-week training follow-up, during the six-week training follow-up, and at a three-month post-training follow-up. The researchers will also be collecting self-report assessments from the participant, observational reports from an Occupational Therapist (OT) and electronic health records to track healthcare utilization and social skills (i.e. communication).
  Interventions: Other: Service Dog Training Program

INTERVENTIONS:
Other: Service Dog Training Program — Participants will spend one hour, two times a week working with professional service dog trainers in order to shape the dog's behavior for it's future role as a service dog for service members with mobility impairments.

SUMMARY:
Preliminary clinical evidence suggests that Service Members with symptoms of post-traumatic stress disorder (PTSD) or Post Traumatic Stress (PTS) who participate in the Service Dog Training Program (SDTP) report improved physical and psychological outcomes, including those with overlapping symptoms associated with traumatic brain injury (TBI) and post-concussion symptoms (PCS).

This study intends to examine the psychological, social, and biological effects of learning how to train a future service dog combined with standard of care for individuals with symptoms of Post-Traumatic Stress (PTS), including those with overlapping TBI and persistent Post-Concussive Symptoms (PCS). Biological, social, and behavioral measures will be collected throughout study participation.

DETAILED DESCRIPTION:
Preliminary clinical evidence suggests that Service Members with symptoms of post-traumatic stress disorder (PTSD) or Post Traumatic Stress (PTS) who participate in the Service Dog Training Program (SDTP) report improved physical and psychological outcomes, including those with overlapping symptoms associated with traumatic brain injury (TBI) and post-concussion symptoms (PCS). Since 2011, over 3,000 injured Service Members have participated in the SDTP. The program entails teaching Service Members how to train service dogs. Participation in this program helps injured Service Members develop skills, such as attention and discipline, which are needed to successfully shape the dog's behavior and are translatable to other social settings. Further, participation in the program appears to enhance the participants' well-being, quality of life, and relationship with significant others, including their children. Moreover, Service Members (SM) who participate in the SDTP report being motivated to participate in the program for the chance of helping other wounded warriors, who will be the recipients of the dogs that they train.

Despite the reported anecdotal benefits from the SDTP, there has been a lack of prospective controlled research studies that examine the efficacy of the program or the biological basis as to how it may be helpful to improve the underlying disease. This study intends to examine the psychological, social, and biological effects of the SDTP combined with standard of care for individuals with symptoms of Post-Traumatic Stress (PTS), including those with overlapping TBI and persistent Post-Concussive Symptoms (PCS). This study will also seek to identify potential psychological, physiological, and/or biological factors that may influence the degree of response from this noninvasive intervention, as well as its potential impact on disease/symptom modification. Further, for those subjects with family members, it will seek to share data with a parallel study ongoing at the University of Maryland to evaluate the effects of the SDTP on family member stress levels, relationship satisfaction, communication evaluate the effects of the SDTP on family member stress levels, relationship satisfaction, communication and parenting.

To accomplish these aims the researchers will recruit DEERS eligible medical beneficiaries who are experiencing PTS and PCS symptoms. Up to 156 participants will be recruited in the National Capital Region (NCR) for a ten-week longitudinal pre-post study, in which each participant will serve as their own control. Additionally, up to 104 participants will be recruited for a three-week longitudinal parallel randomized study will be available for participants recruited through the National Intrepid Center of Excellence (NICoE) 4-week Intensive Outpatient Program (IOP).

Each participant in the active group will train a service dog using methods that facilitate a relationship between the trainer and dog for the gradual shaping of desired behavior. Self-report measures of behavioral symptoms will be given weekly throughout participation in this study. Biological measures, including blood collection, HR, BP, etc. will be collected at baseline, during the three-week training follow-up, during the six-week training follow-up (NCR participants only), and at a three-month post-training followup (optional for NICoE IOP participants). The researchers will also be collecting self-report assessments from the participant, observational reports from an Occupational Therapist (OT) and electronic health records to track healthcare utilization and social skills (i.e. communication).

The study is being carried out in collaboration with the Center for Neuroscience and Regenerative Medicine (CNRM). Under this collaboration, the study will use the CNRM Core Resources including the CNRM Biorepository. Data stored and shared within the CNRM Data Repository will be coded, and upon destruction of the Master List, de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18-65 years old at time of consent.
* Participants must be DEERS eligible men or women from active duty, reserve, National Guard components, retirees, dependents and other Secretarial Designees.
* Participants must have a diagnosis of one of the following:
* PTSD or PTS symptoms (participants must score greater than or equal to 30 on the PCL-5 at screening)
* Anxiety Disorder NOS, Unspecified Trauma Related Disorder, Unspecified Anxiety Disorder, or Adjustment Disorder with evidence of the Service Member experiencing one or more traumatic event (meeting Criterion A of PTSD in DSM 5), and evidence of intrusion symptoms, avoidance symptoms, negative changes in cognitions and mood, and alterations in arousal and reactivity related to the traumatic event or events (Criteria B, C, D, and E of PTSD in DSM 5) persisting beyond 30 days (Criterion F of PTSD in DSM 5)
* Participant may be of any race, ethnicity, or gender.
* Participants with a history of clinician diagnosed TBI are eligible to participate, given the considerable overlap between PTS symptomatology and post-concussive symptoms postacutely.
* Participant must be able to speak and read English, and be able to consent.

Exclusion Criteria:

* Participants must not be younger than 18 years old or other than 65 years old at the time of consent.
* Participant must not show current suicidal/homicidal plans (if the participant expresses current suicidal/homicidal plans, clearance from the participant's current behavioral health team can be provided).
* Participant must not exhibit violent or psychotic behavior.
* Participant must not currently or in the past month have been in an inpatient psychiatric health treatment program.
* Participant must not currently have an active substance abuse disorder or been in a substance abuse program in the past month.
* Participant must not have problems that limit cognitive competency to understand study procedures, including the ability to provide informed consent (e.g., severe TBI). Participant must not be unwilling to answer the study questionnaires.
* Participant must not be afraid of or allergic to dogs.
* Participant cannot be enrolled or participating in any other interventional study for PTS or PTSD treatment.
* Participants cannot currently or in the past six months have participated in clinical service dog training. Clinical service dog training is defined as a type of animal assisted therapy where patients train service dogs as part of a complementary treatment intervention aimed at reducing symptoms associated with physical and psychological injuries. Individuals who have completed a group or individual session in the past six months that only provided an informational overview of the service dog training program will be eligible for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Change in symptom severity using the Post-traumatic Stress Checklist (PCL-5) | The PCL-5 will be collected at screening as part of the inclusion criteria, and subsequently once a week until the end of the 10-week study period, as well as at the 3-month follow-up visit.
  A 20-item self-report measure that assesses changes in symptom severity of PTSD to include, monitoring symptom change during/after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. This instrument will be used for inclusion criteria for the study as well as to assess change during the course of the study.
Change in symptom severity using the Generalized Anxiety Disorder-7 (GAD-7) | The GAD-7 will be collected once a week from start of study until the end of the 10-week study period, as well as at the 3-month follow-up visit.
  A 7-item self-report measure that assesses an individual's level of anxiety from 0 (least severe) to 21 (most severe). The measure has excellent internal consistency (Cronbach alpha = 0.92) and test-retest reliability (intraclass correlation = 0.83). GAD-7 takes less than 5 minutes to complete.
Change in symptom severity using the Patient Health Questionnaire (PHQ-9) | The PHQ-9 will be collected once a week from start of study until the end of the 10-week study period, as well as at the 3-month follow-up visit.
  A 9-item measure of depression from 0 (least severe) to 27 (most severe). The measure has excellent internal reliability (Cronbach's alpha = 0.89), and discriminant validity was supported by ROC analyses that indicated area under the curve for the PHQ-9 in diagnosing depression was 0.095.
Change in symptom severity using the Connor-Davidson Resilience Scale (CD-RISC) | The CD-RISC will be completed at the 4-week, 7-week, 10-week, and 3-month follow-up visits.
  A 25-item self-report measure to help quantify resilience and, as a clinical measure, to assess treatment response on a scale from 0 (least resilient) to 100 (most resilient). The measure has high internal consistency (Cronbach's alpha = 0.89) and test-retest reliability (intra-class correlation = 0.87).
Change in symptom severity using the Defense and Veterans Pain Rating Scale (DVPRS) | The DVPRS will be completed at the 4-week, 7-week, 10-week, and 3-month follow-up visits, as well as after each participant training session (twice a week).
  A visual pain scale to assess individual's pain intensity on a scale of 0-10 (10 being most severe pain), with an additional 4 questions to assess pain's interference with the participant's activity, sleep, mood, and stress.
Change in symptom severity using the Perceived Stress Scale (PSS) | The PSS will be completed at the 4-week, 7-week, 10-week, and 3-month follow-up visits.
  A 10-item measure that assesses an individual's appraisal of their life stressors from 0 (least perceived stress) to 40 (most perceived stress). The PSS demonstrates good reliability (0.84 to 0.86) and face validity, and it is predictive of biological indicators of stress in humans with correlation coefficients ranging from 0.52 to 0.76 for symptomalogical measures.
Change in symptom severity using the Pittsburgh Sleep Quality Index (PSQI) | The PSQI will be completed at the 4-week, 7-week, 10-week, and 3-month follow-up visits.
  A 19-item self-report measure (with 5 additional questions rated by the bedpartner or roommate) evaluating sleep quality and disturbances with lower scores indicating better sleep. The PSQI demonstrates high internal reliability (Cronbach's alpha = 0.83) and test-retest reliability (r = 0.68 to 0.79).
Change in symptom severity using the CDC's Health-related Quality of Life Instrument (HRQOL-14) | The HRQOL-14 will be completed at the 4-week, 7-week, 10-week, and 3-month follow-up visits.
  A 14-item self-report measure that assesses quality of life based on "healthy days" measures and symptoms and activity limitations.
Changes in cortisol | Blood will be collected at baseline (Week 0-1), Week 3, Week 6, and at the 3 month follow-up visit.
  Blood collection not exceeding 40 mL per time point.
Changes in cytokines | Blood will be collected at baseline (Week 0-1), Week 3, Week 6, and at the 3 month follow-up visit.
  Blood collection not exceeding 40 mL per time point. Cytokines strongly associated with PTSD and depression include pro-inflammatory factors IFNG, IL-12, IL-6, and TNF alpha. Cytokines will be measured by multiplex or single immunoassays.
Gene expression | Blood will be collected at baseline for full genome sequencing.
  Blood collection not exceeding 40 mL. DNA genomic variants will be measured by whole genome sequencing.

SECONDARY OUTCOMES:
Changes in scores on Service Dog Training Program (SDTP) Trainer Evaluation Form | The SDTP Trainer Evaluation Form will be completed by the professional dog trainer after each training session, which occurs twice a week from Week 4 through Week 10.
  Questions that will be answered by the dog trainer about the participant. It includes questions about the participant's: level of engagement, ability to understand instruction, ability to communicate instructions praise to the dog, and level of frustration.
Lexington Attachment to Pets Scale (LAPS) | The LAPS will be collected at Week 4.
  A 23-item self-report measure that assesses an individual's attachment to pets with higher scores indicating less attachment to pets. The measure has excellent internal consistency (Cronbach alpha = 0.93).
Life Events Checklist for DSM-5 (LEC-5) | The LEC-5 will be collected at Weeks 4 and 10.
  A 17-item self-report measure designed to screen for potentially traumatic events in an individual's lifetime. The LEC-5 assesses exposure to 16 events known to potentially result in PTSD or distress and includes one additional item assessing any other extraordinarily stressful event not captured in the first 16 items.
Medical Outcome Study - Social Support Survey (MOS-SSS) | The MOS-SSS will be collected at Week 4 and the 3-month follow-up visit.
  A 19-item instrument that assesses perceived social support on a scale from 19 (least social support) to 95 (most social support). The measure is comprised of four support scales, including: emotional/informational, tangible, affectionate, and positive social interaction. The measure has excellent internal consistency (Cronbach alpha = 0.91 to 0.96).
Neurobehavioral Symptom Inventory (NSI) | The NSI will be collected weekly from start of session through the 10-week training period, and again at the 3-month follow-up visit.
  A 22-item measure to assess post-concussive symptoms in individual's who suffered a TBI. The NSI demonstrates high internal consistency (Cronbach's alpha = 0.95).
Pet Attitude Scale (PAS) | The PAS will be collected at the Week 4 visit.
  An 18-item measure to assess human-animal bonding with higher scores indicating a more negative attitude towards pets. The measure has excellent internal consistency (Cronbach alpha = 0.94).
Ohio State University TBI Identification Method - Short Form (OSU-TBI-ID-SF) | The OSU-TBI will be collected at Week 4.
  A structured clinical interview that confirms the diagnosis of mTBI and/or multiple concussion/blast exposures.
Assessment of Communication and Interaction Skill (ACIS) | The ACIS will take place at the start of study, then subsequently every 3 weeks until the end of the 10-week training period. It will be administered once more at the 3-month follow-up visit.
  An observational assessment that gathers data on communication and interaction skills. The ACIS looks at three domains (physicality, information exchange, and relations) and describe different aspects of communication and interaction.
Changes in Heart Rate | Heart rate will take place at all major study visits (Weeks 4, 7, 10, and 3-month follow-up), as well as during each training session twice a week from Week 4 through Week 10.
  Heart rate will be measured using a standard arm cuff.
Changes in Blood Pressure | Blood pressure will take place at all major study visits (Weeks 4, 7, 10, and 3-month follow-up), as well as during each training session twice a week from Week 4 through Week 10.
  Blood pressure will be measured using a standard arm cuff.
Changes in Anthropometric Data measured in inches | Anthropometric data will be collected at Weeks 4, 7, 10, and the 3-month follow-up visit.
  Neck, waist, and hip measurements using inches
Changes in Weight | Weight measurements will be collected at Weeks 4, 7, 10, and the 3-month follow-up visit.
  Weight measured in pounds.
Qualitative Interview | The Qualitative Interview will take place at Week 10 and the 3-month follow-up visit.
  The goal of the qualitative portion of this study is to examine the participants' experience with the SDTP. We are interested in identifying and describing which elements of the intervention are most effective in engaging participants and bringing about behavior change as well as which ones are least effective.
Changes in number of medical visits | Healthcare Utilization Records will be updated during the major study visits at Week 0, Week 4, Week 7, Week 10, and the 3-month follow-up visit.
  Healthcare utilization records will be collected through review of the participants Electronic Health Records (EHR). Study participants will be reviewed for their number of medical visits.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pasquina, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No